CLINICAL TRIAL: NCT05413616
Title: The Effect of a Combined Personalized Nutritional Intervention and a Personalized Graded Activity Functional Training Program on Physical Performance in Hospitalized Older Patients, Compared to Usual Care: A Randomized Clinical Trial
Brief Title: The Effect of a Combined Personalized Nutritional Intervention and a Personalized Graded Activity Functional Training Program on Physical Performance in Hospitalized Older Patients, Compared to Usual Care
Acronym: FITFOOD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-6664
Record Dates: First submitted 2022-05-19; First posted 2022-06-10 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Old Age; Atrophy
Keywords: nutrition; protein; exercise; sarcopenia; older people; vitamin D
MeSH Terms: conditions — Atrophy; Motor Activity; Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention)
- FITFOOD lifestyle intervention (Experimental): Lifestyle intervention consisting of both a nutritional and exercise intervention.
  Interventions: Behavioral: FITFOOD lifestyle intervention

INTERVENTIONS:
Behavioral: FITFOOD lifestyle intervention — Lifestyle intervention with a nutritional and exercise component.
  Arms: FITFOOD lifestyle intervention

SUMMARY:
This project aims to improve physical performance in older patients, by offering a personalized combined nutritional intervention with a physical activity training program. The intervention starts at hospital admittance and is continued after discharge in the home care setting, supported by an e-health application.

DETAILED DESCRIPTION:
Rationale: The older hospitalized population is growing and specifically at risk for decreased muscle mass and physical functioning and has a negative influence on activities of daily living, independence, quality of life, re-admissions, and nursing home placement. Current knowledge shows that a physical activity training programs consisting of tailored resistance and endurance exercise can improve muscle mass in healthy elderly. Nutritional interventions in conjunction with physical activity based on individual protein requirements, high quality protein and timing of protein intake can further stimulate muscle protein synthesis. The effect of a combined nutritional intervention with physical activity in healthy individuals and athletes has been studied before, but not in older hospitalized patients. A personalized combined physical activity program and a nutritional intervention could be a solution and is an exciting emerging field of research with the potential to dramatically improve patient outcomes.

The average hospital admittance is 4 to 5 days in which the prevention of the decline in muscle mass and physical performance can be initiated but not improved. Thus, the translation of a prolonged combined intervention to home care is essential. To support the combined personalized nutritional intervention and physical exercise intervention during hospitalization and home care, an eHealth application for and with older patients can be beneficial.

Objective: This project aims to improve physical performance in older patients, by offering a personalized combined nutritional intervention with a physical activity training program. The intervention starts at hospital admittance, and is continued after discharge in the home care setting, supported by an e-health application.

Study design: The study will be performed as a randomized clinical trial. Study population: The study population hospitalized adult patients of ≥65 years, living in the Nijmegen area within the Radboud University Medical Centre.

Intervention: One group receives a personalized nutritional intervention by a dietician combines with a functional training program by physical therapists. The nutritional intervention focuses on adequate protein intake, type, and timing of protein. The exercise program will make use of goal setting throughout the intervention period to optimize the training effect . The control group will receive usual care.

Study parameters: The primary study outcome is based on the difference in change in physical performance between baseline and after 3 months of intervention of the intervention and the control group (usual care). This will be analyzed using multilevel mixed model corrected by potential confounders, measured by the Timed up & Go test (TUG), a sensitive tool to measure physical performance in elderly.

Secondary: As a secondary outcome, the effect on short physical performance battery, muscle strength, muscle mass, nutritional status, movement, independence, quality of life, clinical outcomes and cost-effectiveness will be studied.

Nature and extent of the burden and risks associated with participation, benefit, and group relatedness: Study measurements are non-invasive. This study will not confer any no additional risks. The intervention will start at hospital admittance and will be continued after discharge in the home setting by a dietician and physiotherapist in their nearby home, which keeps the burden for the patient relatively low and is an extra service for the patient. Protein supplementation will be delivered within the save amounts. Possible serious reactions to the intervention will be noted as SAE's.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥65 years
* Living within the Nijmegen area (within 40km)
* Admitted to clinical ward of Radboudumc or CWZ
* Understanding and speaking of the Dutch language
* Mentally competent
* Signed informed consent

Exclusion Criteria:

* Complete use of tube feeding or parenteral nutrition
* Renal insufficiency (MDRD-GFR < 30ml/min)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2022-07-04 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Timed Up & Go | Baseline, 1 day before hospital release, 4 weeks after baseline, 12 weeks after baseline, 24 weeks after baseline.
  TUG

SECONDARY OUTCOMES:
Change in Short Physical Performance Battery | Baseline, 1 day before hospital release, 4 weeks after baseline, 12 weeks after baseline, 24 weeks after baseline.
  Short Physical Performance Battery (scale: 0-12, a high score indicates no disability, a low score means disabilities may be present or developing).
Change in muscle strength | Baseline, 1 day before hospital release, 12 weeks after baseline, 24 weeks after baseline.
  Handgrip strength
Change in muscle mass | Baseline, 1 day before hospital release, 12 weeks after baseline, 24 weeks after baseline.
  BIA
Change in nutritional status | Baseline, 1 day before hospital release, 4 weeks after baseline, 12 weeks after baseline, 24 weeks after baseline.
  Patient-Generated Subjective Global Assessment (PG-SGA). Scale: 0-49 (low score: no intervention needed. Score>9: serious indication for intervention)
Change in nutritional intake (energy, protein). | Baseline, 1 day before hospital release, 4 weeks after baseline, 12 weeks after baseline, 24 weeks after baseline.
  Food diary.
Change in movement according to actometer | Baseline, 1 day before hospital release, 12 weeks after baseline, 24 weeks after baseline.
  Activ8 measurement will assess movement during 1 week for each measurement point
Change in activities of daily living | Baseline, 1 day before hospital release, 12 weeks after baseline, 24 weeks after baseline.
  LLFDI-CAT (Late-Life Function and Disability Instrument Computer Adaptive Test). LLFDI-CAT scores are transformed to a scale with mean = 50 and standard deviation =10.
  Lower scores correspond to more limitation.
Change in quality of life | Baseline, 1 day before hospital release, 12 weeks after baseline, 24 weeks after baseline.
  EQ-5D-5L (EuroQol 5-level five-dimensional questionnaire). Scores 1-5 where 1 is good and 5 indicates issues or problems.
Clinical outcomes: length of hospital stay | 24 weeks after baseline
  Length of hospital stay
Clinical outcomes: re-admission | 24 weeks after baseline
  Re-admission
Clinical outcomes: complications | 24 weeks after baseline
  Complications
Clinical outcomes: mortality | 24 weeks after baseline
  Mortality
Medical consumption | Baseline
  iMCQ: iMTA Medical Consumption Questionnaire. Medical consumption will be measured using iMCQ and costs are calculated using Dutch reference values.
Medical consumption | 12 weeks after baseline, 24 weeks after baseline
  iMCQ: iMTA Medical Consumption Questionnaire. Medical consumption will be measured using iMCQ and costs are calculated using Dutch reference values.
Risk for Sarcopenia | Baseline, 1 day before hospital release, 4 weeks after baseline, 12 weeks after baseline, 24 weeks after baseline.
  SARC-F: Strength, Assistance with walking, Rise from a chair, Climb stairs (scored 0-1-, higher score means higher risk for sarcopenia) and Falls

CONTACTS AND LOCATIONS:
Locations (1):
- Sabien van Exter, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van Exter SH, Koenders N, van der Wees PJ, Drenth JPH, van den Berg MGA. Lessons learned from a combined, personalized lifestyle intervention in hospitalized patients at risk for sarcopenia: a feasibility study. Disabil Rehabil. 2025 Jul;47(14):3679-3686. doi: 10.1080/09638288.2024.2426685. Epub 2024 Nov 12. PMID 39530465